CLINICAL TRIAL: NCT02512393
Title: Transcranial Direct Current Stimulation in Older Persons With Knee Pain: Randomized Pilot Study
Brief Title: Transcranial Direct Current Stimulation in Older Persons With Knee Pain (Knee Pain and tDCS): Randomized Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: University of Florida (Other)
Responsible Party: Principal Investigator, Hyochol Ahn, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB201500357-2
Record Dates: First submitted 2015-07-29; First posted 2015-07-30 (Estimated); Results first posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active tDCS (Experimental): This group will receive five daily sessions of 2mA, 20 minutes of Transcranial Direct Current Stimulation (tDCS). The anode electrode will be placed over M1 (C3 or C4 according to the 10-20 system for EEG electrode placement) of the hemisphere contralateral to the affected knee, and the cathode electrode will be placed over the supraorbital region (SO) ipsilateral to the affected knee (M1-SO montage). In addition, the following test will performed: X-Rays, Walking Test, Assessment of Physical Performance, Assessment of Sensitivity to Heat, Assessment of Sensitivity to Pressure, Assessment of Sensitivity to Mechanical Stimulation, Assessment of balance, chair stand, and gait speed, Assessment of conditioned pain modulation, and Blood test.
  Interventions: Device: Active tDCS
- Sham tDCS (Sham Comparator): This group will receive five daily sessions of 2mA, current for 30 seconds tDCS. The anode electrode will be placed over M1 (C3 or C4 according to the 10-20 system for EEG electrode placement) of the hemisphere contralateral to the affected knee, and the cathode electrode will be placed over the supraorbital region (SO) ipsilateral to the affected knee (M1-SO montage). In addition, the following test will performed: X-Rays, Walking Test, Assessment of Physical Performance, Assessment of Sensitivity to Heat, Assessment of Sensitivity to Pressure, Assessment of Sensitivity to Mechanical Stimulation, Assessment of balance, chair stand, Assessment of conditioned pain modulation, and gait speed and Blood test.
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Active tDCS — This group will receive tDCS with a constant current of 2 mA intensity will be applied for 20 minutes once a day for five consecutive days using a pair of thick (0.3 cm) rectangular surface sponge electrodes (5 cm x 7 cm) saturated with 10 mL of saline solution. The anode electrode will be placed over M1 (C3 or C4 according to the 10-20 system for EEG electrode placement) of the hemisphere contralateral to the affected knee, and the cathode electrode will be placed over the supraorbital region (SO) ipsilateral to the affected knee (M1-SO montage).
  Other Names: Transcranial Direct Current Stimulation
  Arms: Active tDCS
Device: Sham tDCS — This group will receive tDCS with a constant current of 2 mA intensity will be applied for 30 seconds once a day for five consecutive days using a pair of thick (0.3 cm) rectangular surface sponge electrodes (5 cm x 7 cm) saturated with 10 mL of saline solution. The anode electrode will be placed over M1 (C3 or C4 according to the 10-20 system for EEG electrode placement) of the hemisphere contralateral to the affected knee, and the cathode electrode will be placed over the supraorbital region (SO) ipsilateral to the affected knee (M1-SO montage).
  Arms: Sham tDCS

SUMMARY:
The purpose of this research is to study the effects of Transcranial Direct Current Stimulation (tDCS) on clinical pain, mobility disability, and pain sensitivity to gain a better understanding of the factors that cause pain and disability in people with knee osteoarthritis (OA). In particular, people from different ethnic and racial groups may experience OA pain differently which is why the focus will be on older Asian Americans and non-Hispanic whites. It is important to find a reason for such difference so that a better treatment can be found for all OA patients. In addition, the research study will examine if there is any ethnic differences in pain and mobility disability. The investigator hypothesize that Asian Americans will report greater pain and mobility disability than non-Hispanic whites, and that active tDCS will result in improvement in pain and disability compared to sham tDCS.

DETAILED DESCRIPTION:
If you participate in the study, the following will happen:

Randomized into one of two groups. Which will either receive the full length session of brain stimulation or a much shorter session of brain stimulation. The shorter version of stimulation looks like and is performed in the same way as the longer electrical stimulation session, but stimulation is stopped before it can have much of an effect on the brain. You will not know which group you have been assigned to while participating in the research, but you may find out at the completion of the research study.

X-Rays will be done on both knees while standing up.

Questionnaires about arthritis pain you are having, your thoughts and feelings about it, and any stress that you may have experienced.

Walking Test will be performed on a flat surface for 6 minutes at a fast pace without help from an assistive device (cane or walker) or another person.

Assessment of Physical Performance requires walking at short distance (about 13 feet), stand up from a chair 5 times without using your arms, and stand in 3 different positions while keeping your balance.

Assessment of Sensitivity to Heat. Heat pain sensitivity will be tested using a commercially available thermal sensory testing machine (Medoc, Inc.) used widely in clinical settings. This machine has a small (about 1 inch by 1 inch) square piece that is used to apply heat to the skin. Heat will be applied to the knees and arms. The amount of heat is controlled by a computer. One or more of the following types of heat stimuli will be delivered: 1) a slowly increasing heat that can be stopped by pressing a button when it becomes warm, painful, or intolerable; 2) a series of 5-10 heat pulses that are brief (less than 2 seconds in duration), and rate how painful each heat pulse feels; and 3) a few longer heat pulses (15-30 seconds) at different temperatures to rate how painful each heat pulse feels. The procedures can be stop at any time.

Assessment of Sensitivity to Pressure will be done using a handheld device with a small rubber tip to apply pressure to the knee, thigh, and shoulder.

Assessment of Sensitivity to Mechanical Stimulation will be done using a handheld probe that has a small nylon tip to tap both the knee and hand.

Blood Draw: Blood will be taken at the baseline visit and at the last visit.

Brain Stimulation: The stimulation technique called transcranial direct current stimulation (tDCS) and it involves placing two sponge-like electrodes on your head and delivering a very weak electrical current to your scalp, which is generated by a 9 volt battery.

In addition, weekly phone calls will be done for the next 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* they have self-reported unilateral or bilateral knee OA pain according to American College of Rheumatology criteria
* they can understand, speak and read English
* they are able to walk for 6-minutes
* they are willing to be randomized to either the intervention or control group
* they are available for five consecutive daily sessions and for a follow-up phone interview each week for three weeks post-stimulation sessions
* they have no plan to change medication regimens for pain throughout the trial
* they are willing and able to provide written informed consent

Exclusion Criteria:

* knee replacement or non-arthroscopic surgery to the affected knee
* serious medical illness, such as uncontrolled hypertension (i.e., Systolic Blood Pressure/Diastolic Blood Pressure of ≥ 150/95), congestive heart failure, pacemaker, or history of acute myocardial infarction
* peripheral neuropathy
* systemic rheumatic disorders, including rheumatoid arthritis, systemic lupus erythematosus, and fibromyalgia
* alcohol/substance abuse
* cognitive impairment (i.e., Mini-Mental Status Exam score ≤ 23)
* history of brain surgery, tumor, seizure, stroke, or intracranial metal implantation
* pregnancy or lactation for females
* hospitalization within the preceding year due to psychiatric illness

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-11; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hyochol Ahn, PhD, ARNP, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- University of Texas Health Science Center at Houston, Houston, Texas, United States

REFERENCES:
- [Derived] Ahn H, Woods AJ, Kunik ME, Bhattacharjee A, Chen Z, Choi E, Fillingim RB. Efficacy of transcranial direct current stimulation over primary motor cortex (anode) and contralateral supraorbital area (cathode) on clinical pain severity and mobility performance in persons with knee osteoarthritis: An experimenter- and participant-blinded, randomized, sham-controlled pilot clinical study. Brain Stimul. 2017 Sep-Oct;10(5):902-909. doi: 10.1016/j.brs.2017.05.007. Epub 2017 May 19. PMID 28566193

RESULTS

PARTICIPANT FLOW:
Groups:
- Active tDCS: This group will receive five daily sessions of 2mA, 20 minutes of Transcranial Direct Current Stimulation (tDCS). The anode electrode will be placed over M1 (C3 or C4 according to the 10-20 system for EEG electrode placement) of the hemisphere contralateral to the affected knee, and the cathode electrode will be placed over the supraorbital region (SO) ipsilateral to the affected knee (M1-SO montage).
- Sham tDCS: This group will receive five daily sessions of 2mA, current for 30 seconds tDCS. The anode electrode will be placed over M1 (C3 or C4 according to the 10-20 system for EEG electrode placement) of the hemisphere contralateral to the affected knee, and the cathode electrode will be placed over the supraorbital region (SO) ipsilateral to the affected knee (M1-SO montage).
Period: Overall Study
Arm/Group | Active tDCS | Sham tDCS
Started | 21 | 20
Completed | 20 | 20
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active tDCS | Sham tDCS | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.60 (9.80) | 59.30 (8.60) | 59.95 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 10 | 9 | 19
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Numeric Rating Scale (NRS) for Pain
Description: Numeric Rating Scale for pain is an 101-point scale for patient self-reporting of pain on a scale of 0 to 100, with 0 being no pain at all and 100 being the worst pain imaginable. The higher the score the worse the pain.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
units on a scale | 27.25 (3.35) | 19.00 (1.72)

2. Primary Outcome: Numeric Rating Scale (NRS) for Pain
Description: as for outcome 1
Time Frame: day 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
units on a scale | 8.75 (1.54) | 12.55 (2.98)

3. Primary Outcome: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale
Description: This is a index to rate the activity of pain, stiffness, and physical function based on a scale of difficulty: 0 = None, 1 = Mild, 2 = Moderate, 3 = Severe, 4 = Extreme; subscales are added up for a summation score. The higher the score, the worse the pain.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
units on a scale | 29.30 (3.68) | 20.40 (2.13)

4. Primary Outcome: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale
Description: as for outcome 3
Time Frame: day 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
units on a scale | 24.20 (2.57) | 19.50 (2.93)

5. Primary Outcome: Short-Form McGill Pain Questionnaire-2 (SF-MPQ-2) Continuous Pain Subscale
Description: This is a questionnaire to rate the pain intensity and related symptoms on a scale of 0 to 10, with 0 being none and 10 being the worst possible. The higher the score the worse the pain.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
units on a scale | 2.25 (0.48) | 1.50 (0.23)

6. Primary Outcome: Short-Form McGill Pain Questionnaire-2 (SF-MPQ-2) Continuous Pain Subscale
Description: as for outcome 5
Time Frame: day 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
units on a scale | 1.29 (0.22) | 1.60 (0.41)

7. Primary Outcome: Short-Form McGill Pain Questionnaire-2 (SF-MPQ-2) Intermittent Pain Subscale
Description: as for outcome 5
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
units on a scale | 1.75 (0.58) | 0.98 (0.28)

8. Primary Outcome: Short-Form McGill Pain Questionnaire-2 (SF-MPQ-2) Intermittent Pain Subscale
Description: This is a index to rate the activity of pain based on a scale of difficulty: 0 = None, 1 = Mild, 2 = Moderate, 3 = Severe, 4 = Extreme. The higher the score, the worse the pain.
Time Frame: day 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
units on a scale | 0.96 (0.33) | 1.15 (0.39)

9. Primary Outcome: Short-Form McGill Pain Questionnaire-2 (SF-MPQ-2) Neuropathic Pain Subscale
Description: as for outcome 5
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
units on a scale | 0.93 (0.29) | 0.80 (0.20)

10. Primary Outcome: Short-Form McGill Pain Questionnaire-2 (SF-MPQ-2) Neuropathic Pain Subscale
Description: as for outcome 5
Time Frame: day 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
units on a scale | 0.54 (0.13) | 0.66 (0.20)

11. Primary Outcome: Short-Form McGill Pain Questionnaire-2 (SF-MPQ-2) Affective Pain Subscale
Description: as for outcome 5
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
units on a scale | 1.58 (0.51) | 0.66 (0.20)

12. Primary Outcome: Short-Form McGill Pain Questionnaire-2 (SF-MPQ-2) Affective Pain Subscale
Description: as for outcome 5
Time Frame: day 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
units on a scale | 0.61 (0.15) | 0.77 (0.21)

13. Primary Outcome: Six-minute Walk Test
Description: The six-minute walk test (6MWT) measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes. The individual is allowed to self-pace and rest as needed as they traverse back and forth along a marked walkway. The lower the score the worse the condition.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
meters | 478.18 (16.46) | 490.71 (18.26)

14. Primary Outcome: Six-minute Walk Test
Description: as for outcome 13
Time Frame: day 5
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
meters | 497.47 (16.75) | 494.26 (18.77)

15. Primary Outcome: Short Physical Performance Battery (SPPB)
Description: This is a group of measures that combines the results of the gait speed, chair stand, and balance tests. The score ranges from 0 (worst performance) to 12 (best performance).
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
units on a scale | 11.05 (0.27) | 11.10 (0.33)

16. Primary Outcome: Short Physical Performance Battery (SPPB)
Description: as for outcome 15
Time Frame: day 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
units on a scale | 11.25 (0.28) | 11.05 (0.33)

17. Primary Outcome: Heat Pain Threshold
Description: Quantitative Sensory Testing (QST) by using heat pain delivered by using thermal probe on the skin.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
Celsius | 41.84 (4.38) | 40.51 (4.69)

18. Primary Outcome: Heat Pain Threshold
Description: Quantitative Sensory Testing (QST) by using heat pain delivered by using thermal probe on the skin.
Time Frame: day 5
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
Celsius | 42.62 (3.20) | 40.18 (4.34)

19. Primary Outcome: Heat Pain Tolerance
Description: Quantitative Sensory Testing (QST) by using heat pain delivered by using thermal probe on the skin.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
Celsius | 46.47 (3.01) | 45.04 (3.59)

20. Primary Outcome: Heat Pain Tolerance
Description: Quantitative Sensory Testing (QST) by using heat pain delivered by using thermal probe on the skin.
Time Frame: day 5
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
Celsius | 47.07 (2.26) | 45.42 (3.50)

21. Primary Outcome: Pressure Pain Threshold
Description: Quantitative Sensory Testing (QST) by using pressure pain delivered by a hand-held algometer.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: kilopascal (kPa)
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
kilopascal (kPa) | 2.61 (1.13) | 2.63 (1.30)

22. Primary Outcome: Pressure Pain Threshold
Description: Quantitative Sensory Testing (QST) by using pressure pain delivered by a hand-held algometer.
Time Frame: day 5
Measure: Mean (Standard Deviation); unit: kilopascal (kPa)
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
kilopascal (kPa) | 3.21 (1.08) | 2.98 (1.10)

23. Primary Outcome: Punctate Mechanical Pain Sensitivity
Description: Quantitative Sensory Testing (QST) by using punctate mechanical pain delivered by a calibrated nylon monofilament.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: kilopascal (kPa)
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
kilopascal (kPa) | 45.85 (31.94) | 46.60 (25.99)

24. Primary Outcome: Punctate Mechanical Pain Sensitivity
Description: Quantitative Sensory Testing (QST) by using punctate mechanical pain delivered by a calibrated nylon monofilament.
Time Frame: day 5
Measure: Mean (Standard Deviation); unit: kilopascal (kPa)
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
kilopascal (kPa) | 42.23 (26.87) | 50.73 (33.61)

25. Primary Outcome: Conditioned Pain Modulation (CPM)
Description: Conditioned pain modulation (CPM) will be done by using a cold pressor procedure on the skin. The measure is scored on a scale, which ranges from zero to infinity. A higher CPM score indicates higher pain inhibition.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
units on a scale | 0.84 (0.69) | 0.73 (0.48)

26. Primary Outcome: Conditioned Pain Modulation (CPM)
Description: as for outcome 25
Time Frame: day 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
units on a scale | 0.94 (0.52) | 0.70 (0.71)

27. Secondary Outcome: Endorphin Level
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
ng/mL | 0.04 (0.01) | 0.04 (0.02)

28. Other Pre Specified Outcome: NIH PROMIS-cognition Will be Compared Between the Two Groups for a Change Between Baseline and Day 5
Description: A score of 50 is the average and a score of 60 is better than average. A score of 40 is the worse score.
Time Frame: Change from baseline and day 5
Reporting Status: Not Posted

29. Other Pre Specified Outcome: Safety Questionnaire Will be Compared Between the Two Groups for a Change Between Baseline, 1, 2, 3, 4, and 5 Days.
Description: This is a questionnaire to assess the presence and severity of adverse events such as headache, tingling, itching, and fatigue, on a scale of 0 to 10, with 0 being not at all and 10 being a highest degree.
Time Frame: Change from baseline, 1, 2, 3, 4, and 5 days
Reporting Status: Not Posted

30. Other Pre Specified Outcome: Coping Strategies Questionnaire-Revised Will be Compared Between the Two Groups for a Change Between Baseline and Day 5
Description: This is a questionnaire to assess pain coping strategies, such as distancing from pain, using a 7-point scale that ranges from never do that to always do that. The higher the scale the greater use.
Time Frame: Change from baseline and day 5
Reporting Status: Not Posted

31. Other Pre Specified Outcome: Positive and Negative Affect Scale Will be Compared Between the Two Groups for a Change Between Baseline and Day 5
Description: This is a questionnaire using a 5-point scale that ranges from very slightly or not at all to extremely. The lower the scale the negative the affect and the higher the scare the positive the affect.
Time Frame: Change from baseline and day 5
Reporting Status: Not Posted

32. Other Pre Specified Outcome: Pain Attitudes Questionnaire-Revised Will be Compared Between the Two Groups for a Change Between Baseline and Day 5
Description: This is a questionnaire to assess pain attitudes, such as stoicism, using a 5-point scale that ranges from strongly disagree to strongly agree. The higher the scale the more stoic.
Time Frame: Change from baseline and day 5
Reporting Status: Not Posted

33. Secondary Outcome: Endorphin Level
Time Frame: day 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
ng/mL | 0.04 (0.02) | 0.05 (0.02)

34. Secondary Outcome: Cortisol Level
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
pg/mL | 47085.48 (36657.95) | 39358.75 (29387.62)

35. Secondary Outcome: Cortisol Level
Time Frame: day 5
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
pg/mL | 46588.50 (32249.18) | 38853.23 (24343.37)

36. Secondary Outcome: C-reactive Protein (CRP) Level
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
ng/mL | 1394.33 (1278.41) | 1758.26 (2833.17)

37. Secondary Outcome: C-reactive Protein (CRP) Level
Time Frame: day 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
ng/mL | 1496.74 (1469.79) | 3372.98 (5490.50)

38. Secondary Outcome: Tumor Necrosis Factor (TNF) Level
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
pg/mL | 7.63 (3.42) | 10.20 (5.78)

39. Secondary Outcome: Tumor Necrosis Factor (TNF) Level
Time Frame: day 5
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
pg/mL | 7.41 (3.27) | 10.36 (5.98)

40. Secondary Outcome: Interleukin 6 (IL-6) Level
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
pg/mL | 2.12 (1.78) | 3.57 (3.65)

41. Secondary Outcome: Interleukin 6 (IL-6) Level
Time Frame: day 5
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
pg/mL | 2.40 (1.43) | 3.37 (2.62)

42. Secondary Outcome: Interleukin 10 (IL-10) Level
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
pg/mL | 6.25 (3.20) | 8.91 (5.36)

43. Secondary Outcome: Interleukin 10 (IL-10) Level
Time Frame: day 5
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20
pg/mL | 5.68 (2.85) | 8.17 (4.56)

ADVERSE EVENTS:
Arm/Group | Active tDCS | Sham tDCS
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes